CLINICAL TRIAL: NCT00173706
Title: Evaluation of the Effects of L-Carnitine Injection in Patients Undergoing Hemodialysis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 930404
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2006-03-01 (Estimated); Status verified 2005-08

CONDITIONS: Cardiac Complications; Signs and Symptoms; Muscle Weakness; Anemia; Hypotension
Keywords: L-Carnitine; hemodialysis; cardiac complications; impaired exercise and functional capacities; muscle symptoms; intradialytic hypotension; erythropoietin-resistant anemia
MeSH Terms: conditions — Signs and Symptoms; Muscle Weakness; Anemia; Hypotension | interventions — Carnitine

INTERVENTIONS:
Drug: L-Carnitine Injection

SUMMARY:
This is a study designed to test the hypothesis that treatment with L-carnitine will improve the quality of life and some specific symptoms and signs in patients with renal failure submitted to hemodialysis.

DETAILED DESCRIPTION:
L-Carnitine is a naturally occurring compound that facilitates the transport of fatty acids into mitochondria for beta-oxidation. A lack of carnitine in hemodialysis patients is caused by insufficient carnitine synthesis and particularly by the loss through dialytic membranes, leading in some patients to carnitine depletion with a relative increase of esterified forms. Many studies have shown that L-carnitine supplementation leads to improvements in several complications seen in uremic patients, including cardiac complications, impaired exercise and functional capacities, muscle symptoms, increased symptomatic intradialytic hypotension, and erythropoietin-resistant anemia, normalizing the reduced carnitine palmitoyl transferase activity in red cells.

ELIGIBILITY:
Inclusion Criteria:

Patients with the following criteria will be eligible for participation in this study:

1. Male or female adults over 18 years of age
2. On hemodialysis for at least one year
3. Interdialysis weight gain < 5%
4. Bicarbonate dialysis 3 times per week
5. Modality of dialysis unchanged for 3 months prior to entry into the study (concerning dialysis-time and mode: bicarbonate, acetate dialysis)
6. Have one of the following symptoms and signs that have not responded to diet or pharmacological intervention:

   1. persistent weakness affecting daily life
   2. malnutrition
   3. anemia (hemoglobin [Hb] < 12 g/dl; hematocrit [Hct] < 30%)
   4. experiencing intradialytic complications (cramping, muscular pain, hypotension, hypertension, head-ache)
7. On regular treatment with vitamin B12 and folates
8. Normal iron status (ferritin > 100 ng/ml; transferrin saturation [TSAT] > 20%)
9. Informed consent obtained
10. Patients with diabetes mellitus are allowed to enter the study if they have stable glycaemic control on diet or pharmacological treatment.

Exclusion Criteria:

Patients displaying one or more of the following criteria will not be eligible for participation in this study:

1. Severe uncontrolled hypertension (systolic > 170; diastolic > 115) outside of dialysis
2. Some patients have echocardiogram (ECHO) defined chronic heart failure. Patients with New York Heart Association (NYHA) class II and class III can be admitted. Patients with class IV must be excluded. Some patients have angina. Patients with stable effort angina well controlled by treatment can be recruited. Absolute exclusion for angina at rest.
3. Major hepatic diseases - chronic active (aggressive) hepatitis or cirrhosis
4. Systemic haematological diseases and tumours
5. Uncontrollable diabetes
6. History of drug and alcohol abuse
7. Positive screening for HIV antibodies
8. Life expectancy of less than one year
9. Uncontrolled hyperparathyroidism (patients with stable bone status can be recruited)
10. Use of immunodepressants during the preceding 4 weeks
11. Changes in corticoid therapy in the preceding 4 weeks
12. Use of experimental drugs during the preceding 4 months
13. Use of L-carnitine during the preceding 4 months
14. Informed consent not obtained
15. Pregnancy
16. Patients already included in other clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-10

PRIMARY OUTCOMES:
weakness
improvement of hypotension and hematology profile
reduction of erythropoietin requirement
increase of plasma carnitine concentration

SECONDARY OUTCOMES:
including all the components of the primary endpoints for their further assessment
improvement of the nutritional indexes
intradialytic complications (muscle symptoms, dyspnea, palpitations)
quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Kwan-Dun Wu, Ph.D, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan